CLINICAL TRIAL: NCT05650268
Title: Effects of Stoss Therapy of Vitamin D3 on Peri-operative Outcomes in Patients Receiving General Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Because of impact from COVID-19 pandemic
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201808006RIPC
Record Dates: First submitted 2021-07-26; First posted 2022-12-14 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2021-08

CONDITIONS: Vitamin D Deficiency; Surgery
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D3 (Experimental): The experimental group will receive 576000 IU in single oral dose of liquid vitamin D3~7 days prior to the surgery.
  Interventions: Drug: Vitamin D3
- Control group (Placebo Comparator): The control group will receive 95% MCT D3~7 days prior to the surgery.
  Interventions: Other: 95% MCT

INTERVENTIONS:
Drug: Vitamin D3 — Receiving 576000 international units in single oral dose of liquid vitamin D 3~7 days prior to the surgery.
  Other Names: Vitamin D
  Arms: Vitamin D3
Other: 95% MCT — 95% MCT supplement 3-7 day before surgery
  Arms: Control group

SUMMARY:
To investigate whether preoperative supplement with high-dose vitamin D3 can reduce the perioperative risk and enhance recovery

DETAILED DESCRIPTION:
Perioperative management for risk reduction in patients undergoing major surgery are taken increasingly important nowadays. The patient factor (age and comorbidities mainly), type of surgery and extent of tissue injury are major contributions to the development perioperative complications. From nutrition support to nutrition therapy, a comprehensive nutrition plays a pivotal role to optimize the above three key factors and hence reduce the perioperative risk. Vitamin D, a pleiotropic hormone with extensive physiological effect, is one of the nutrients critical to perioperative outcomes. It not only meets the essential demand of surgical patients, such as wound care, infection control, metabolic support and organ support, but also attenuates oxidative stress, modulates dys-inflammation and repair the damaged organelles like telomere and mitochondria. This is a double-blind, randomized controlled trial in a single center. Sixty eligible adult patients who will undergo general surgery are to be included.

The experimental group will receive 576000 IU in single oral dose of liquid vitamin D 3~7 days prior to the surgery. The primary endpoint is rapid recovery index, such as bowel recovery, pain control, sedation and fatigue assessment. The secondary endpoints include perioperative inflammatory indexes, hemodynamic parameters, glycemic control as well as safety evaluation of vitamin D.

ELIGIBILITY:
Inclusion Criteria:

* 20 years or older
* Adult patients who will receive general surgery

Exclusion Criteria:

* Chronic liver diseases
* Hypercalcemia
* Using estrogen drug, bisphosphonate, other durgs to treat bone diseases
* Sarcoidosis, Multiple myeloma or Primary hyperparathyroidism
* Pregnant women
* Other trial participation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Mortality rate | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Yin-Yi Han, MD,PhD, Principal Investigator — National Taiwan University Hospital

IPD SHARING:
Plan to Share IPD: No